CLINICAL TRIAL: NCT00618748
Title: Safety and Efficacy of Olanzapine (LY170053) in the Long-term Treatment for Patients With Bipolar I Disorder, Depressed
Brief Title: Safety and Efficacy of Olanzapine in the Long-term Treatment for Bipolar I Disorder, Depressed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11682; F1D-JE-HGMS (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-Olanzapine (Experimental): Participants who received olanzapine 5-20 mg/day in Study HGMP (NCT#00510146), received olanzapine 5-20 mg/day, orally for 24 weeks.
  Interventions: Drug: Olanzapine
- Pre-Placebo (Experimental): Participants who received placebo in acute phase of Study HGMP (NCT#00510146), received olanzapine 5-20 mg/day, orally for 24 weeks.
  Interventions: Drug: Olanzapine
- New Olanzapine (Experimental): Participants who did not participate in Study HGMP (NCT#00510146), received olanzapine 5-20 mg/day, orally for 48 weeks.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 5-20 mg/day, oral, daily
  Other Names: LY170053

SUMMARY:
To assess the efficacy and safety of olanzapine in the long-term treatment for patients with bipolar I disorder, depressed.

DETAILED DESCRIPTION:
This is an open-label, multi-center, long-term treatment study conducted only in Japanese sites. The subjects are patients who fulfill the diagnostic criteria for bipolar I disorder, most recent episode depressed, as defined in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) (296.50=unspecified, 296.52=moderate severity, 296.53=severe without psychotic features, 296.54=severe with psychotic features), who have completed Study HGMP (NCT#00510146) and patients who did not participate in Study HGMP who have been recruited to participate in Study HGMS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged 18 to less than 75 years.
2. Each patient must be reliable, have a level of understanding sufficient to perform all tests and examinations required by the protocol, and must understand the nature of the study and have provided informed consent.
3. All female patients must test negative for pregnancy.
4. Females of breast-feeding potential must agree not to breastfeed an infant during the study and for 1 month following the last dose of study drug.
5. Male patients who are not surgically sterilized must agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
6. Patients must fulfill the diagnostic criteria for bipolar I disorder, most recent episode depressed, as defined in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR).
7. Patients must have experienced, in the opinion of the investigator, at least one previous manic or mixed episode, as defined in the DSM-IV-TR.
8. Patients must have a current Young Mania Rating Scale (YMRS) Total score =<8.

Exclusion Criteria:

1. Is investigator site personnel directly affiliated with this study or their immediate families.
2. Is a Lilly employee.
3. Has previously completed or withdrawn from this study or any other study investigating olanzapine.
4. Is pregnant or nursing.
5. Has a serious, unstable illness such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4599) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

REFERENCES:
- [Derived] Katagiri H, Tohen M, McDonnell DP, Fujikoshi S, Case M, Kanba S, Takahashi M, Gomez JC. Safety and efficacy of olanzapine in the long-term treatment of Japanese patients with bipolar I disorder, depression: an integrated analysis. Psychiatry Clin Neurosci. 2014 Jul;68(7):498-505. doi: 10.1111/pcn.12156. Epub 2014 Mar 4. PMID 24417745
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Olanzapine: Participants who received olanzapine in Study HGMP (NCT#00510146), received olanzapine 5-20 mg/day, orally for 24 weeks.
Period: Overall Study
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Started | 56 | 25 | 20
Completed | 45 | 20 | 6
Not Completed | 11 | 5 | 14
Not completed — Adverse Event | 4 | 3 | 8
Not completed — Physician Decision | 3 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine | Total
Number analyzed (Participants) | 56 | 25 | 20 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 39.31 (10.48) | 37.53 (7.64) | 39.13 (9.56) | 38.84 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 14 | 13 | 61
  Male | 22 | 11 | 7 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  East Asian | 56 | 25 | 20 | 101
Region of Enrollment [Number; unit: participants]
  Japan | 56 | 25 | 20 | 101
Montgomery- Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  units on a scale | 8.05 (7.50) | 9.72 (6.48) | 16.45 (9.03) | 10.13 (8.18)
Young Mania Rating Scale (YMRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
  units on a scale | 0.38 (1.10) | 0.40 (0.76) | 0.45 (0.83) | 0.40 (0.97)
Clinical Global Improvement- Bipolar (CGI-BP) - Mania [Mean (Standard Deviation); unit: units on a scale] — CGI-BP is a measure of illness severity especially adapted for bipolar illness. It allows rating of mania, depression, and overall illness. The Mania score ranges from 1 (normal, not ill) to 7 (very seriously ill).
  units on a scale | 1.09 (0.35) | 1.00 (0.00) | 1.00 (0.00) | 1.05 (0.26)
CGI-BP - Depression [Mean (Standard Deviation); unit: units on a scale] — CGI-BP is a measure of illness severity especially adapted for bipolar illness. It allows rating of mania, depression, and overall illness. The Depression score ranges from 1 (normal, not ill) to 7 (very seriously ill).
  units on a scale | 2.23 (0.95) | 2.48 (0.82) | 3.55 (1.15) | 2.55 (1.08)
CGI-BP - Overall [Mean (Standard Deviation); unit: units on a scale] — CGI-BP is a measure of illness severity especially adapted for bipolar illness. It allows rating of mania, depression, and overall illness. The Overall Illness score ranges from 1 (normal, not ill) to 7 (very seriously ill).
  units on a scale | 2.20 (0.92) | 2.40 (0.82) | 3.25 (1.02) | 2.46 (1.00)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation
Description: An adverse event (AE) is an untoward medical event associated with the use of the study drug or study procedure, whether or not it is considered related to the study drug or study procedure. Results presented are the percentage of participants who experienced an adverse event that resulted in the discontinuation of the study.
Time Frame: Baseline through 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: All randomized Participants.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
percentage of participants | 7.1 | 12.0 | 40.0

2. Secondary Outcome: Change From Baseline in Glucose and Lipid Panel at Week 24 or Week 48 Endpoint
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit result.
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
millimole/Liter
  Glucose, Fasting | 0.03 (0.47) | 0.37 (0.55) | 0.68 (1.31)
  Cholesterol | 0.033 (0.699) | 0.040 (0.716) | 0.086 (1.031)
  Low-density lipoprotein ( LDL) Cholesterol | 0.141 (0.676) | -0.034 (0.731) | 0.008 (0.855)
  High-density lipoprotein ( HDL) Cholesterol | -0.036 (0.221) | -0.046 (0.212) | -0.074 (0.239)
  Triglycerides | -0.108 (0.543) | 0.485 (1.415) | 0.382 (1.270)

3. Secondary Outcome: Change From Baseline in Weight at Week 24 or Week 48 Endpoint
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit result.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
kilograms | 0.29 (2.79) | 0.92 (3.02) | 5.36 (4.34)

4. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 24 or Week 48 Endpoint
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and at least one non-missing post baseline value, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
units on a scale | -0.2 (8.3) | -0.4 (6.5) | -5.8 (11.6)

5. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Week 24 or Week 48 Endpoint
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
units on a scale | 0.4 (1.5) | -0.2 (1.0) | -0.1 (1.7)

6. Secondary Outcome: Change From Baseline in Clinical Global Improvement- Bipolar (CGI-BP) at Week 24 or Week 48 Endpoint
Description: CGI-BP is a measure of illness severity especially adapted for bipolar illness. It allows rating of mania, depression, and overall illness. The scores for mania, depression, and overall illness each range from 1 (normal, not ill) to 7 (very seriously ill).
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
units on a scale
  CGI-BP Mania | -0.1 (0.4) | 0.1 (0.3) | 0.1 (0.2)
  CGI-BP Depression | -0.3 (0.9) | -0.0 (0.9) | -1.1 (1.3)
  CGI-BP Overall Bipolar Illness | -0.3 (1.0) | -0.1 (0.7) | -0.9 (1.1)

7. Secondary Outcome: Percentage of Participants With Emergence of Mania at Week 24 or Week 48
Description: Emergence of mania is defined as first occurrence of score of >=15 in the YMRS total score in the post-baseline period of Acute Phase. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: All Randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
percentage of participants | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With High Suicidality at Week 24 or Week 48
Description: The MINI module C (MINI-C) is a rating scale for severity of suicidal thoughts and behaviors. The MINI-C is composed of 12 Yes/No questions with variable scores assigned to each question. The scale ranges from 0 to 52 with higher scores indicating a greater presence of suicidal thoughts and/or behaviors. Based upon scores, suicidality is defined as Low (1-8), Medium (9-16), and High (>=17).
Time Frame: 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit value.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
percentage of participants | 3.6 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Extra-Pyramidal Symptoms (EPS) at Week 24 or Week 48
Description: EPS symptoms measured by DIEPSS are grouped into 4 categories: Parkinsonism, akathisia, dystonia, and dyskinesia. Severity ranges from level 0 (none, normal) to 4 (severe). A participant is deemed to have EPS at endpoint if they have an abnormal endpoint. Normal baseline Parkinsonism is defined as a score not ≥3 on 1 item or ≥2 on 2 items; abnormal endpoint is a score ≥3 on 1 item or ≥2 on 2 items, or an increase of 3 on Parkinsonism total. Normal baseline akathisia, dystonia and dyskinesia is defined as a score <2; abnormal endpoint is a score ≥2 or an increase ≥2 from that baseline score.
Time Frame: 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with a normal baseline and an endpoint result. For Parkinsonism, normal baseline is defined as a score not ≥3 on 1 item or ≥2 on 2 items. Normal baseline akathisia, dystonia and dyskinesia is defined as a score <2.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
percentage of participants
  Akathisia | 0 | 0 | 0
  Dyskinesia | 0 | 0 | 0
  Dystonia | 0 | 0 | 0
  Parkinsonism | 3.6 | 0 | 5.0

10. Secondary Outcome: Change From Baseline in Hemoglobin (HbA1c) at Week 24 or Week 48 Endpoint
Description: HbA1c is a test that measures the amount of glycated hemoglobin in the blood over prolonged periods of time.
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit result.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
percentage of glycated hemoglobin | -0.016 (0.259) | 0.036 (0.243) | 0.180 (0.282)

11. Secondary Outcome: Change From Baseline in Prolactin at Week 24 or Week 48 Endpoint
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit result.
Measure: Mean (Standard Deviation); unit: microgram/Liter
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 25 | 20
microgram/Liter | -1.669 (10.498) | -0.388 (14.179) | 3.383 (18.731)

12. Secondary Outcome: Change From Baseline to in QTcF at Week 24 or Week 48 Endpoint
Description: Time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole, fixed correction factor (QTcF interval)
Time Frame: baseline, 24 weeks (pre-olanzapine and pre-placebo) or 48 weeks (new olanzapine)
Population: Participants with non-missing baseline value and the specified visit result.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Number analyzed (Participants) | 56 | 24 | 20
millisecond (msec) | -1.7 (16.6) | -8.5 (13.1) | -3.4 (13.9)

ADVERSE EVENTS:
Arm/Group | Pre-Olanzapine | Pre-Placebo | New Olanzapine
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/25 | 1/20
Other Adverse Events (participants affected / at risk) | 34/56 | 13/25 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Olanzapine (N=56) | Pre-Placebo (N=25) | New Olanzapine (N=20)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Olanzapine (N=56) | Pre-Placebo (N=25) | New Olanzapine (N=20)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperprolactinaemia (Endocrine disorders) | 3 (5) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (9) | 1 (1) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 4 (5)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood prolactin increased (Investigations) | 4 (4) | 1 (1) | 0 (0)
Blood triglycerides decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 3 (3) | 1 (1) | 14 (15)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 5 (6)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days